CLINICAL TRIAL: NCT02615119
Title: Neural Basis of Meal Related Interoceptive Dysfunction in Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017-002
Record Dates: First submitted 2015-11-18; First posted 2015-11-26 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Anorexia Nervosa; Major Depressive Disorder; Generalized Anxiety Disorder; Panic Disorder; Brain Injury
Keywords: heartbeat; respiration; interoception; anxiety; eating
MeSH Terms: conditions — Anorexia Nervosa; Depressive Disorder, Major; Generalized Anxiety Disorder; Panic Disorder; Brain Injuries; Respiratory Aspiration; Anxiety Disorders | interventions — Isoproterenol; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Anorexia nervosa (Experimental): Intravenous bolus infusions of isoproterenol (up to 4 micrograms per infusion) and normal saline.
  Interventions: Drug: Isoproterenol; Drug: Normal saline
- Generalized anxiety disorder (Experimental): Intravenous bolus infusions of isoproterenol (up to 4 micrograms per infusion) and normal saline.
  Interventions: Drug: Isoproterenol; Drug: Normal saline
- Panic disorder (Experimental): Intravenous bolus infusions of isoproterenol (up to 4 micrograms per infusion) and normal saline.
  Interventions: Drug: Isoproterenol; Drug: Normal saline
- Major depressive disorder (Experimental): Intravenous bolus infusions of isoproterenol (up to 4 micrograms per infusion) and normal saline.
  Interventions: Drug: Isoproterenol; Drug: Normal saline
- Brain injury (Experimental): Intravenous bolus infusions of isoproterenol (up to 4 micrograms per infusion) and normal saline.
  Interventions: Drug: Isoproterenol; Drug: Normal saline
- Healthy comparison (Active Comparator): Intravenous bolus infusions of isoproterenol (up to 4 micrograms per infusion) and normal saline.
  Interventions: Drug: Isoproterenol; Drug: Normal saline

INTERVENTIONS:
Drug: Isoproterenol — Intravenous infusions of isoproterenol, delivered in a randomized double blinded order, in each participant from each group. Participants will rate the experience of heartbeat and breathing sensations as well as anxiety induced by the infusion.
  Other Names: Isuprel
Drug: Normal saline — Intravenous infusions of normal saline, delivered in a randomized double blinded order, in each participant from each group. Participants will rate the experience of heartbeat and breathing sensations as well as anxiety induced by the infusion.
  Other Names: Saline

SUMMARY:
This study aims to identify the brain regions responsible for encoding cardiorespiratory 'interoceptive' sensations and determine whether they are dysfunctional in individuals affected by eating disorders, anxiety, depression, or brain injury. By evaluating the same interoceptive sensations across different human illnesses, the investigators hope to provide convergent evidence resulting in identification of core underlying neural processes, and to discern relative contributions in each condition.

DETAILED DESCRIPTION:
The human brain has constant access to a multitude of complex signals, which it must simplify and organize in order to sustain the integrity of the organism. Many of these signals originate from outside of the body, such as lights, sounds, and smells, and much is known about how humans consciously perceive these 'exteroceptive' signals and how the human brain represents them. Comparatively little is known about how the human brain processes 'interoceptive' signals originating from inside of the body, despite the fact that the brain has access to far more of them (for instance, intestinal tension, bladder distension, breath, heartbeat, body temperature, blood pressure, serum osmolality, inflammation, proprioception etc.).

The current study study therefore aims to identify the brain regions responsible for encoding cardiorespiratory 'interoceptive' sensations and determine whether they are dysfunctional in individuals affected by eating disorders, anxiety, depression, or brain injury. Participants in this study will receive stimulation of the cardiorespiratory channel of the interoceptive system using bolus intravenous infusions of isoproterenol, a peripherally acting medication similar to adrenaline, and saline. Stimulation will occur during functional magnetic resonance imaging (fMRI) as well as outside of the fMRI scanner. After the scan participants will consume a meal. By evaluating the same interoceptive sensations across different human illnesses, the investigators hope to provide convergent evidence resulting in identification of core underlying neural processes, and to discern relative contributions in each condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual 5 (DSM 5) criteria for anorexia nervosa and age 18 to 40, or generalized anxiety disorder, or panic disorder, or major depressive disorder, or brain injury caused either by herpes simplex encephalitis or Urbach-Wiethe disease.

Exclusion Criteria:

* DSM 5 diagnosis with any of the following: Schizophrenia spectrum and other psychotic disorders, bipolar and related disorders, antisocial personality disorder, active suicidal ideation with intent or plan
* Current cardiac arrhythmia
* Current respiratory disease
* Seizure disorder
* MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/ wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a professional metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60-120 minutes; prior neurosurgery; tattoos or cosmetic makeup with metal dyes, unwillingness to remove body piercings, and pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Change in cardiorespiratory sensation intensity | Baseline
  Visual analogue rating of intensity of heartbeat and breathing sensations (scale: 0 to 10) through study completion (e.g., the day of testing).

SECONDARY OUTCOMES:
Change in anxiety level | Baseline
  Visual analog rating of level of anxiety (scale: 0 to 10) through study completion, an average of 2 weeks.
Generalized anxiety disorder severity (Generalized Anxiety Disorder 7 scale) | Baseline
  7 questions on anxiety symptoms
Panic disorder severity (Panic Disorder Severity scale) | Baseline
  panic symptoms questionnaire
Major depressive disorder severity (Patient Health Questionnaire-9 scale) | Baseline
  9 questions on depression symptoms
Eating disorder severity (Eating Disorder Examination scale) | Baseline
  questionnaire about eating disorder symptoms

OTHER OUTCOMES:
Resting cardiac interoceptive sensitivity (heartbeat tapping task tap latencies (in milliseconds)) | Baseline
  subject taps with their finger their own perceived heart beat
Systolic and diastolic blood pressure (millimeters of mercury; mmHg) during the autonomic task of the valsalva maneuver | Baseline
  blood pressure assessed
Systolic and diastolic blood pressure (millimeters of mercury; mmHg) during the autonomic handgrip task. | Baseline
  blood pressure assessed
Systolic and diastolic blood pressure (millimeters of mercury; mmHg) during the autonomic task of mental arithmetic. | Baseline
  blood pressure assessed
Systolic and diastolic blood pressure (millimeters of mercury; mmHg) during the autonomic cold pressor task. | Baseline
  blood pressure assessed
Systolic and diastolic blood pressure (millimeters of mercury; mmHg) during the autonomic task of breath holding). | Baseline
  blood pressure assessed
Structural magnetic resonance imaging (cortical thickness in millimeters cubed). | Baseline
  Structural MRI measure: cortical thickness.
Functional magnetic resonance imaging (Blood Oxygenation Level Dependent i.e. BOLD signal) | Baseline
  Functional MRI measure: task based activation change
EEG (coherence in alpha, beta, theta, delta, gamma frequencies, in Hertz (Hz)) | Baseline
  EEG: global and local coherence.
Change in heart rate | Baseline
  Average heart rate change versus pre-infusion baseline
Change in breathing pattern | Baseline
  Average respiratory volume variability change versus pre-infusion baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sahib S Khalsa, MD, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teed AR, Feinstein JS, Puhl M, Lapidus RC, Upshaw V, Kuplicki RT, Bodurka J, Ajijola OA, Kaye WH, Thompson WK, Paulus MP, Khalsa SS. Association of Generalized Anxiety Disorder With Autonomic Hypersensitivity and Blunted Ventromedial Prefrontal Cortex Activity During Peripheral Adrenergic Stimulation: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Apr 1;79(4):323-332. doi: 10.1001/jamapsychiatry.2021.4225. PMID 35107563

DOCUMENTS (1):
  • Informed Consent Form (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT02615119/ICF_000.pdf